CLINICAL TRIAL: NCT02299908
Title: Ultrasound-guided Transverses Abdominis Plane Block in Inguinal Herniorrhaphy: Randomized Controlled Clinical Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Patricia Salazar Villegas (Other)
Responsible Party: Sponsor-Investigator, Patricia Salazar Villegas, Master in Business Administration, Universidad de Caldas
Organization: Universidad de Caldas (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VIP 1691514
Record Dates: First submitted 2014-11-17; First posted 2014-11-24 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Pain, Postoperative
Keywords: Hernia, Inguinal; Herniorrhaphy; Abdominal Wall; Analgesia; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative; Hernia, Inguinal; Agnosia | interventions — Anesthesia, Local; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAP block with Bupivacaine at 0.25% (Experimental): Intervention: Injection of local anesthetics in the transverses abdominal plane
  Interventions: Drug: TAP block with Bupivacaine at 0.25%
- Placebo saline solution (Placebo Comparator): Placebo: Injection of saline solution in the transverses abdominal plane
  Interventions: Drug: Placebo saline solution

INTERVENTIONS:
Drug: TAP block with Bupivacaine at 0.25% — Application of 20 mL of local anesthetic bupivacaine at 0.25% in the transverse abdominis plane (TAP) under ultrasound guidance. This area (TAP) is between the anterior fascia of the transverse abdominal muscle and the posterior fascia of the internal oblique muscle, through which the thoracic nerve fibers and a portion of the first lumbar pass. This intervention will be done 10 minutes before conducting the ipsilateral inguinal herniorrhaphy in a single application.
  Other Names: TAP block; Infiltration of local anesthetic; Local anesthesia in inguinal herniorrhaphy
  Arms: TAP block with Bupivacaine at 0.25%
Drug: Placebo saline solution — Application of 20 mL of saline solution in the transverse abdominis plane (TAP).
  Other Names: Saline solution
  Arms: Placebo saline solution

SUMMARY:
Acute postoperative pain is one of the most important centers of therapeutic attention in postoperative phase of any procedure. It is a complex entity that requires a multiple intervention to be treated and, depending on the intervened surgical site, it has different approaches.

Despite attempts to reduce postoperative pain by implementing management protocols, rates of pain prevalence from moderate acute to severe pain are still reported as high as 50% in the first 24 postoperative hours. Among the surgeries that report greater intensity of postoperative pain is open inguinal Herniorrhaphy. That is why several techniques have been described for the management of acute pain in this surgery postoperative, among which PAT blocking has shown to be beneficial in some studies. However, some reports question its usefulness but with the emergence of ultrasound-guided techniques for its realization, interest in this blockage has grown back.

This study aims to demonstrate the utility of the PAT blocking in the management of acute pain of pre-peritoneal inguinal herniorrhaphy with mesh.

DETAILED DESCRIPTION:
1. Patient registry:

The cases will be recorded by an external agent who will verify compliance with the protocol by the treating physicians (surgeons and anesthesiologists); additionally this agent will interview patients for the processing of the instrument and will also collect the proper information of the procedure. At random and in an unannounced way, visits will be made to the centers of attention to verify that the procedure was done according to what had been agreed.

Additionally when the full record of the patients is registered in a database, they will be called one by one to confirm the information collected. Further records are sought in the systematized medical history in order to verify additional information.

a. Quality assurance plan: i. Each record will be completed by an external agent to the surgical procedure who will be trained for this work according to the methodological design of the study.

ii. Regular visits are made to the information collection site to confirm compliance with attention and randomization protocols.

iii. Information collected on the instrument will be confirmed with each patient's the clinical history.

b. Data verification for range and consistency: i. Each of the instruments for each unit of analysis will be typed in a database by the same person (who will be trained in the methodological design of the study) who will monitor that each variable has been collected according to the categories previously established for that variable.

ii. One second revision of the database will be carried out by one of the researchers who will review column by column categories, so that they are consistent with the predefined rules for that range: Additionally, compatibility between these categories and other categories of variables that must be compatible will be verified. For example, the hour of completion of surgery is later than the start time, etc.

c. Verification of data for Accuracy, Completeness and Representativeness i. Each instrument collected will be verified, with surgical description carried out by the surgeon, anesthesia report made by the anesthesiologist and medical developments made by the hospital physician in charge of patient care in the postoperative period. In case of finding any inconsistency, the confirmation of the information will proceed through an additional call to the patient and the treating specialists if necessary.

ii. Record of the patient's inclusion in the protocol of the clinical trial, guiding the treating physicians in the active pursuit of the variables under study, will be included in all electronic medical records.

d. Data Dictionary:

* Consecutive: Unique number for each unit of analysis. Source: Patient. Code: Does not apply. Ranges: 1, 2, 3, 4, 5, and so on. Type: Organization.
* Date: Day, month and year in which the surgery is carried out. Source: Medical history. Code: Does not apply. Ranges: Day: 1 a 31. Month: 1 a 12, Year: 2015. Type: Organization.
* Age: Age at time of surgery. Source: Identification Number. Code: Does not apply. Ranges: 18, 19, 20, and so on. Type: Base.
* Sex: Gender. Source: Patient. Code: Does not apply. Ranges: Male, Female. Type: Base.
* Social Stratum: Economic level. Source: Patient. Code: Does not apply. Ranges: 1, 2, 3, 4, 5, 6. Type: Base.
* Education: Educational level. Source: Patient. Code: Does not apply. Ranges: None, Primary School, Secondary School, technical, technological, professional, specialist, Master's, Doctoral degree. Type: Base.
* Laterality: Side of hernia. Source: Patient. Code: Does not apply. Ranges: Right, Left. Type: Base.
* ASA: Surgical risk. Source: Medical history. Code: Does not apply. Ranges: 1, 2, 3, 4, 5. Type: Clinic.
* Weight: Weight in kilograms. Source: Medical history. Code: Does not apply. Ranges: 30, 31, 32, and so on. Type: Base.
* Height: Height in meters. Source: Medical history. Code: Does not apply. Ranges: 1.4, 1.41, 1,42, and so on. Type: Base.
* Background: Diseases that the patient has. Source: Medical history and patient. Code: Does not apply. Ranges: Asthma, chronic obstructive pulmonary disease (COPD), hypertension, diabetes, heart failure, etc. Type: Clinic.
* Lockout duration: Block performance time (minutes). Source: Surgery room. Code: Does not apply. Ranges: 2, 3, 4, 5, and so on. Type: Anesthetic.
* Duration of surgery: Surgery completion time (minutes). Source: Surgery room. Code: Does not apply. Ranges: 15, 16, 17, and so on. Type: Surgical.
* Adverse Reactions: Side effects and complications. Source: Surgery room. Code: Does not apply. Ranges: Hypotension, bradycardia, arrhythmias, aspiration of blood, viscera perforation, hematoma, femoral nerve block, infiltration resistance. Type: Primary result.
* Realization: Specialist who performed the lock. Source: Surgery room. Code: Does not apply. Ranges: 1, 2. Type: Anesthetic.
* Pain 1: Visual Analog Scale (VAS) when anesthetic medication suspended. Source: Patient. Code: Does not apply. Ranges: 1, 2, 3, 4, 5, 6, 7, 8, 9, 10. Type: Primary result.
* Rescue 1: Number of rescue doses of morphine applied early after anesthetics have been suspended. Source: Recovery nurse. Code: Does not apply. Ranges: 1, 2, 3, 4, and so on. Type: Secondary result.
* Adverse effect 1: Adverse effect presented early after anesthetics is suspended. Source: Recovery nurse. Code: Does not apply. Ranges: Vomiting, nausea, itching, dry mouth, drowsiness, respiratory depression, none, other. Type: Secondary result.
* Pain 2: VAS 24 hours after anesthetic medication is suspended. Source: Patient. Code: Does not apply. Ranges: 1, 2, 3, 4, 5, 6, 7, 8, 9, 10. Type: Primary result.
* Rescue 2: Number of rescue tramadol dosage applied between the first hour and 24-hour after anesthetic is suspended. Source: Patient. Code: Does not apply. Ranges: 1, 2, 3, 4, and so on. Type: Secondary result.
* Adverse effect 2: Adverse effect occurred between first hour and 24-hours after anesthetic is suspended. Source: Patient. Code: Does not apply. Ranges: Vomiting, nausea, itching, dry mouth, drowsiness, respiratory depression, none, other. Type: Secondary result.
* Intervention: Application of local PAT anesthetic. Source: Currency format (Randomization). Code: Does not apply. Ranges: Yes (Intervention), No (Placebo). Type: Intervention.

  e. Standard Operation Procedures: i. Registration operation:
  1. Patient Recruitment:

     1. All patients scheduled for inguinal herniorrhaphy by the surgeon, will be reported by the administrative programming group to the researchers who will attend the preoperative evaluation by anesthesiology to practice informed consent and inclusion and exclusion criteria. Patients that can continue with the protocol will be included in the study.
     2. The day of the surgery the surgical instrumentation group will perform the patients' randomization with a consecutive (identification number) and, without knowing the patient, will take to the operating room the substance to apply in the PAT.
  2. Data collection:

     1. During surgery a research assistant who is blind to the applied substance, shall record the data collection instrument based on what he observes in the operating room and on what he questions in the first hour after the suspension of anesthetics in the post-anesthesia care room.
     2. After 24 hours of suspending the anesthetic, the research assistant will call the patient to question him about the necessary information to complete the data collection instrument of.
  3. Data management:

     1. The missing information in the database will be completed through review of medical records, interview with the surgeon, anesthesiologist and unit post-anesthesia care nurse. The information still needed, will be supplemented through a call to the patient. If despite the above it is not possible to get the required information, the case will be withdrawn for further analysis by intention to treat.
     2. Visits, audits and random checks to confirm the effectiveness of the data collection will be made.

     ii. Analysis Activities:

  <!-- -->

  1. Data analysis:

     Information of the instruments will be typed for the development of a database which will be complemented by the intervention variable the day determined to collect the sample. After that it will be delivered to the researchers who will undertake the analysis and interpretation so that later they can make the socialization of results.
  2. Adverse effects report:

     Whenever an adverse outcome is evidenced, it will be reported to the researchers and treating physicians (surgeon and anesthesiologist). Additionally the patient will be informed. Likewise it will be notified on clinical trial data base.
  3. Change management:

     1. If it is necessary to make a change to the protocol or data collection, researchers will meet to discuss the best option which does not affect the overall outcome of the investigation, but also which does not put in an additional hazard the patients' safety. When this aspect is defined a statement to the entire group of research will be issued.
     2. If a severe and frequent adverse reaction occurs, the possibility to suspend the controlled clinical trial will be determined between the researchers and the medical ethics committee.

     f. Evaluation of the sample size:

     i. Number of participants: The sample size was calculated using the formula for mean difference in analytical studies with a confidence index of 95%, a margin of error of 5%, a statistical power of 80%, a variance of 10% and a minimum differential detection value of 2.8%, compared to which a sample of 40 patients was obtained. With a loss rate of 10% the sample size was expanded to 44 patients.

     ii. Years participated: Since it is an acute pain study 24 hours were determined to monitor.

     g. Missing data plan:

     i. Missing data will be completed with clinical history, interview o professionals involved with patient care, calls and / or visits to patients. If data loss remains an analysis by intention to treat will proceed.

     h. Statistic analysis plan: i. Frequency distribution and qualitative variables association tables will be made, statistical significance for p values less than 0.05 will be determined, association between intervention variable and primary outcome and secondary outcome variables will be sought using for t his purpose the statistics analysis plan.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years attending Servicios Especiales de Salud (SES) Hospital of Caldas and Santa Sofia Hospital for inguinal hernia surgery.
* Physical status classification of the American Society of Anesthesiologists (ASA) (ASA I: healthy patient with no history or comorbidity and ASA II patients with compensated systemic disease).
* Acceptance to complete the informed consent.

Exclusion Criteria:

* Bilateral inguinal hernia.
* Allergy to drugs used in the study protocol (propofol, remifentanil, dipyrone, Dexamethasone, Tramadol, Morphine, Bupivacaine, Cephalexin, Cefazolin, Lidocaine, Sevoflurane, Chlorhexidine, Adrenaline, Naproxen, Acetaminophen)
* Lack of communication with the patient
* Inadequate social support network and interaction with the physician.
* Spinal Anesthesia
* Herniorrhaphy without mesh.
* Pregnancy
* Abuse of psychoactive substances.
* Daily consumption of opioids.
* Consumption of analgesics during the last 24 hours prior to surgery.
* Infection at the incision site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-07 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Postoperative acute pain measured by the visual analog scale (VAS) from 1-10 with 1 being the lowest and 10 the highest intensity after one hour of anesthesia suspension. | 1 hour after the suspension of anesthesia

SECONDARY OUTCOMES:
Opioid Consumption 1 | 1 hour after the suspension of anesthesia
  Number of rescue doses of 2 mg of Morphine each one, used for pain management in the first hour after stopping the administration of anesthetic agents
Adverse reactions 1 | 1 hour after the suspension of anesthesia
  Adverse reactions present in the first hour after the suspension of anesthesia
Postoperative acute pain 2 | 24 hours after the suspension of anesthesia
Adverse reactions 2 | 24 hours after the suspension of anesthesia
Opioid Consumption 2 | 24 hours after the suspension of anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Oscar D Aguirre Ospina, Specialist, Principal Investigator — Universidad de Caldas
Locations (2):
- Colombia (2):
  - Hospital Departamental Universitario Santa Sofía de Caldas, Manizales, Caldas Department
  - SES Hospital de Caldas, Manizales, Caldas Department